CLINICAL TRIAL: NCT06246578
Title: Concordance of Hypoglycemia Measurement in People With Type 1 Diabetes, With Simultaneous Use of Two Devices for Continuous Glucose Measurement: Abbott Freestyle Libre 2 and Dexcom G7
Brief Title: Concordance of Hypoglycemia Measurement With Simultaneous Use of Two Devices for Continuous Glucose Measurement.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recent published work comparing different sensors has outdated our study. It is meaningless to continue to compare "old" sensors, which are updated to never version with different performance.
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Klavs Würgler Hansen, Professor, Central Jutland Regional Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 791575
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Hypoglycemia; Continuous glucose monitoring; Dexcom; Libre; Blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Comparison of nearly simultaneous interstitial glucose values obtained by Dexcom G 7 and Libre 2 sensors for continuous glucose monitoring and blood glucose measured with Contour Next one
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Within patient comparison (Other): Simultaneous glucose measurement with Libre 2 sensor and Contour Next One in patients using Dexcom G7
  Interventions: Device: Continuos glucose monitoring and blood glucose measurement

INTERVENTIONS:
Device: Continuos glucose monitoring and blood glucose measurement — The individuals who use Dexcom G 7 sensors for continous glucose monitoring is in addition applied a Libre 2 sensor and asked to wear both sensors for 14 days. In case of a Dexcom glucose value < 5 mmol/l, the participants is aked to measure a blood glucose as well uising fingerprick and Contour Next One

SUMMARY:
The aim of this study is to compare two frequently used sensors for continuous glucose monitoring (CGM); Freestyle Libre and Dexcom G 7. More precisely, the investigators want to investigate if there is any difference in the hypoglycemic range for these two devices.

DETAILED DESCRIPTION:
The investigators are including adults with type 1 diabetes who already are using a Dexcom G 7, in their diabetes treatment. Simultaneously with their Dexcom G7, the participants will get the Libre 2 sensor attached, and are to wear this for a period of 14 days. The Libre sensor is a Freetsyle Libre 2. Glucose data are compared for paired values within a time interval of 5 min or less. In this way the investigators have access to nearly simultaneous glucose values from two different CGM's. In addition, the participants are given a Contour Next One, and are asked to measure their blood glukose with fingerprick if their Dexcom registers a glucose value < 5 mmol/l.

By this project, we hope to gain more precise information about the two most widely distributed CGMs, and their function in the hypoglycemic area. This, can have impact on healthcare professionals' future therapeutic instructions, regarding the use of insulin adjustment and carbohydrate compensation.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes Using Dexcom G 7 -

Exclusion Criteria:

Do not want to participate

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference between paired blood glucose values and simultaneous Dexcom and Libre glucose values | 5 minutes or less between the glucose values compared
  Difference between paired blood glucose values and simultaneous CGM values for Dexcom and Libre for Dexcom values < 5 mmol/l
Difference between paired Dexcom and Libre glucose values | 5 minutes or less between the glucose values compared
  Difference between paired simultaneous CGM value for Dexcom and Libre for all measured glucose values.

CONTACTS AND LOCATIONS:
Overall Officials: Klavs W Hansen, MD, Study Director — Silkeborg Regional Hospital
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Date, time and glucose values
Time Frame: At time of submitting the manuscript
Access Criteria: on reasonable request